CLINICAL TRIAL: NCT05074134
Title: An Open Label Phase 1 Study in Healthy Adult Male Subjects to Investigate the Absorption, Metabolism, and Excretion of [14C]-TNP-2092 Following a Single Intravenous Dose Administration
Brief Title: Absorption, Metabolism, and Excretion Study of [14C]-TNP-2092
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TenNor Therapeutics Limited (Industry)
Responsible Party: Sponsor
Organization: TenNor Therapeutics Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TNP-2092-IV-08
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]-TNP-2092 (Experimental)
  Interventions: Drug: [14C]-TNP-2092

INTERVENTIONS:
Drug: [14C]-TNP-2092 — Subjects will receive a single intravenous (IV) dose of 300 mg/3 µCi [14C]-TNP-2092 administered over 60 minutes (± 10 minutes).

SUMMARY:
This is an open-label, single dose, Phase 1 study conducted at a single study center in the United States (USA). This study will evaluate the absorption, metabolism and elimination (AME), mass balance, safety and tolerability of a single dose of intravenously administered [14C]-TNP-2092.

Healthy men aged 18 to 55, will be screened, and subjects who meet all eligibility criteria and provide written informed consent will be enrolled into the study within 28 days of Screening.

Subjects will be admitted to the clinical unit on the day prior to dosing (Day -1). Subjects will fast overnight and then given a standard breakfast 30 min prior to dosing.

Six subjects will be enrolled in the study and each will receive a single intravenous (IV) dose of 300 mg/3 μCi [14C]-TNP-2092 administered over 60 minutes (±10 minutes).

DETAILED DESCRIPTION:
This is an open-label, single dose, Phase 1 study conducted at a single study center in the United States (USA). This study will evaluate the absorption, metabolism and elimination (AME), mass balance, safety and tolerability of a single dose of intravenously administered [14C]-TNP-2092 Healthy men aged 18 to 55, will be screened, and subjects who meet all eligibility criteria and provide written informed consent will be enrolled into the study within 28 days of Screening.

Subjects will be admitted to the clinical unit on the day prior to dosing (Day 1). Subjects will fast overnight and then given a standard breakfast 30 min prior to dosing.

Six subjects will be enrolled in the study and each will receive a single intravenous (IV) dose of 300 mg/3 µCi [14C]-TNP-2092 administered over 60 minutes (±10 minutes).

Subjects will remain in the unit for 7 days after dosing (until morning of Day 8) for observation and collection of whole blood, urine and fecal samples.

Whole blood samples will be collected at pre-dose (-30 minutes) and at 15 minutes, 30 minutes, 45 minutes, 1 h (end of infusion), and at 1 h 5 minutes, 1 h 10 minutes, 1 h 15 minutes, 1 h 30 minutes, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours after initiation of the [14C]-TNP-2092 infusion (n=25 timepoints per subject). Depending on 14C radiolabel recovery, an additional whole blood sample may be collected on Day 15 (336 hours after initiation dosing) for a total of n=26 timepoints per subject. These samples will be used to determine concentrations of TNP-2092 (in plasma), metabolite profiling (in plasma), and total [14C] (whole blood and plasma).

Urine will be continuously collected for [14C] recovery, and metabolite assessments from the time of admission until immediately prior to dosing (pre dose) and over the following collection intervals: 0-8, 8-16, 16-24, 24-48, 48-72, 72-96, 96-120, 120-144 and 144-168 hours (Day 8) after initiation of the [14C]-TNP 2092 infusion (n=10 timepoints per subject). Depending on 14C radiolabel recovery, additional urine samples may be collected on Days 14 and 15 (312-336 hours after dosing).

Feces will be continuously collected for metabolite and [14C] recovery assessments from the time of admission until immediately prior to dosing (pre dose) and over the following collection intervals: 0-24, 24-48, 48-72, 72-96, 96-120, 120-144 and 144-168 hours (Day 8) after initiation of the [14C]-TNP-2092 infusion (n=8 timepoints per subject). Depending on 14C radiolabel recovery, additional fecal samples may be collected on Days 14 and 15 (312-336 hours after dosing).

Safety will be assessed by physical examination, vital signs (VS), 12-lead electrocardiograms, clinical laboratory tests (serum chemistry panel, hematology, coagulation, and urinalysis), use of concomitant medications, collection of adverse events, and by unscheduled assessments as needed for management of adverse events.

Subjects will be discharged from the CPC on Day 8 after completion of all 168h timepoint assessments. The Investigator will indicate whether ≥90% of the 14C radiolabel has been recovered in samples collected through 168h; if so, Day 8 will be the final study visit. If recovery of 14C in excreta is <90% by the time of discharge on Day 8, subjects will return to the site for an additional 24-hour PK confinement period on Days 14-15 (312-336h). The date of study completion for each subject will be defined as the last day that PK samples are collected. To avoid enrolling a participant with systemic 14C excess, samples of urine and/or blood (either whole blood or plasma) obtained at Screening must show no significant excess of 14C over environmental background level.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of understanding the written informed consent form (ICF), willingly provide valid, signed written informed consent, and willing and able to comply with the schedule, requirements, and restrictions of the study
2. Males between 18 and 55 years of age (inclusive) at the time of Screening
3. Body mass index (BMI) ≥18.0 kg/m2 and ≤32.0 kg/m2 at Screening; body weight ≥55.0 kg and ≤100.0 kg at Screening
4. Considered to be in good health by the Investigator, as determined by medical history, physical examination, VS measurements, 12-lead ECG, and clinical laboratory test results
5. Male subjects with female sexual partner(s) of reproductive potential may be enrolled if the male:

   1. is documented to be surgically sterile (i.e., successfully vasectomized), or
   2. agrees to use 2 methods of highly effective contraception and agree to refrain from sperm donation from the time of Screening through 90 days post dose
6. Negative serology results for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), and human immunodeficiency virus antibody (HIV Ab)
7. Non-smoker (with no use of other tobacco or nicotine containing products, in any form), as documented by history (no nicotine within 6 months prior to Screening) and a negative cotinine test at Screening and Admission See Section 5.3 for details of nicotine and tobacco restrictions
8. Negative results for drugs of abuse and alcohol at Screening and Admission
9. Content of 14C in urine, whole blood, and/or plasma (per Investigator discretion) samples obtained at Screening does not significantly exceed the general environmental background 14C level At present, background level of 14C is 104 percent Modern Carbon (pMC). To be eligible for study enrollment, subjects must have ≤30 pMC in a plasma or urine sample analyzed with sodium benzoate carbon carrier or ≤150 pMC for a sample analyzed directly (with no carbon carrier).
10. Willing to comply with Pharmaron's COVID-19 policies.

Exclusion Criteria:

1. Any contraindication to the use of rifampin/rifamycin or a fluoroquinolone
2. History or presence of any condition (e.g., chronic diarrhea) or prior surgery (e.g., gastric bypass) that, in the opinion of the Investigator, poses a significant risk to subject safety and/or achievement of study objectives
3. Clinically significant abnormal medical history, or any abnormal findings on physical examination, VS, ECG, or laboratory tests at Screening, Admission, or pre dose on Day 1 that, in the opinion of the Investigator, could jeopardize achieving the study objectives and/or compromise the subject's safety
4. History of cancer that has not been in full remission for >5 years (except basal cell skin cancer or squamous cell skin cancer with history of curative treatment and no recurrence for >1 year prior to Screening), as judged by the Investigator
5. Acute illness within 14 days prior to study drug administration on Day 1, unless mild in severity and enrollment is approved by both the Investigator and Sponsor's medical representative
6. COVID-19 positive for active disease
7. Any history of allergic drug reactions
8. History or presence of alcohol or drug abuse within 2 years prior to Screening
9. Recent history of incomplete bladder emptying with voiding or awakening more than once at night to void
10. Usual habit of <1 or >3 bowel movements per day
11. Exposure to radiation for therapeutic or diagnostic reasons (except dental X rays and plain X rays of thorax and bony skeleton) within the past 12 months prior to study drug administration on Day 1, or worker occupationally exposed to radiation
12. Participation in another clinical study in which a [14C] labeled drug was administered within 1 year prior to Admission
13. Administration of another investigational medication within 30 days (or 5 half lives, whichever is longer) prior to study drug administration
14. Participation in an investigational device study within 30 days prior to study drug administration
15. Any ECG abnormality considered to be clinically significant by the Investigator
16. QTcF interval (QT interval corrected for heart rate per Fridericia's formula) >450 msec at Screening, Admission, or pre dose on Day 1
17. Family history of long QT syndrome or of unexplained sudden death in a first-degree relative under 50 years of age
18. Documented congenital or acquired long QT syndrome
19. Glomerular filtration rate (GFR) ≤80 mL/min/1.73 m2, as estimated by the Chronic Kidney Disease Epidemiology Collaboration (CKD EPI) equation
20. Presence of clinically significant hypertension, defined as systolic blood pressure (SBP) >140 mmHg and/or diastolic blood pressure (DBP) >90 mmHg, at Screening or Admission
21. Presence of clinically significant hypotension, defined as SBP <90 mmHg and/or DBP <50 mmHg, at Screening or Admission
22. Loss or donation of blood (approximately 500 mL) within 60 days prior to study drug administration on Day 1; donation of bone marrow or peripheral stem cells within 90 days prior to study drug administration on Day 1; or donation of plasma within 30 days prior to study drug administration on Day 1
23. Excessive consumption of alcohol, defined as >3 alcoholic beverages per day (12 ounces of beer [354 mL], 5 ounces of wine [148 mL] or 1.5 ounce of distilled spirits [44 mL] is approximately equivalent to 1 alcoholic beverage)
24. Excessive consumption of coffee, tea, cola or other caffeinated beverages; excessive consumption is defined as >6 servings per day (1 serving contains approximately 120 mg caffeine)
25. Venous access considered inadequate for PK sample collection; history or evidence of adverse symptoms associated with phlebotomy or blood donation
26. Employee or family member of the Investigator, study site personnel or Sponsor
27. Use/consumption of any medications or substances listed as prohibited
28. Any other reason that, in the opinion of the Investigator, would render the subject unsuitable for study enrollment.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2021-10-16 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Mass balance of TNP-2092 and the percentages of radiolabel recovered in urine and feces | Day 7
  Percent (%) for each radiolabeled drug-related material will be determined in plasma,urine and feces.
Pharmacokinetics (PK) of TNP-2092 in plasma | Day 7
  AUC(Area under the plasma concentration) will be determined, using Linear/Log trapezoidal method, from plasma concentration data for TNP-2092
Pharmacokinetics (PK) of TNP-2092 in plasma | Day 7
  t1/2 (apparent terminal elimination half life) will be estimated for TNP-2092 from the terminal portion of its plasma concentration versus time plot

SECONDARY OUTCOMES:
Routes and rates of elimination of [14C] TNP 2092 | Day 7
  Recovery (as % administered dose) of total radioactivity in urine and feces.

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmaron Clinical Pharmacology Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No